CLINICAL TRIAL: NCT04341090
Title: A Randomized, Open-label, Single Dose, Three-period, Six-sequences, Crossover Study of High-fat and Low-fat Meal Effect on the Pharmacokinetics of Apatinib Mesylate in Chinese Healthy Adult Subjects
Brief Title: A Food Effect Study of Apatinib Mesylate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HR-APTN-I-009
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Experimental): Drug:apatinib mesylate tablet , 250 mg, 3 discrete single doses separated by 4-days: the first dose will be after fasted, the second dose will be after low-fat meal, the third dose will be after high-fat meal
  Interventions: Drug: Apatinib Mesylate
- Arm 2 (Experimental): Drug:apatinib mesylate tablet , 250 mg, 3 discrete single doses separated by 4-days: the first dose will be after high-fat meal, the second dose will be after fasted, the third dose will be after low-fat meal
  Interventions: Drug: Apatinib Mesylate
- Arm 3 (Experimental): Drug:apatinib mesylate tablet , 250 mg, 3 discrete single doses separated by 4-days: the first dose will be after low-fat meal, the second dose will be after high-fat meal, the third dose will be after fasted
  Interventions: Drug: Apatinib Mesylate
- Arm 4 (Experimental): Drug:apatinib mesylate tablet , 250 mg, 3 discrete single doses separated by 4-days: the first dose will be after fasted, the second dose will be after high-fat meal, the third dose will be after low-fat meal
  Interventions: Drug: Apatinib Mesylate
- Arm 5 (Experimental): Drug:apatinib mesylate tablet , 250 mg, 3 discrete single doses separated by 4-days: the first dose will be after low-fat meal, the second dose will be after fasted, the third dose will be after high-fat meal
  Interventions: Drug: Apatinib Mesylate
- Arm 6 (Experimental): Drug:apatinib mesylate tablet , 250 mg, 3 discrete single doses separated by 4-days: the first dose will be after high-fat meal, the second dose will be after low-fat meal, the third dose will be after fasted
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — Single dose of apatinib mesylate after high-fat meal, low fat meal and fast

SUMMARY:
The primary objective of the study was to assess the effect of high-fat and low-fat meal on the pharmacokinetics of apatinib mesylate in Chinese adult healthy subjects.

The secondary objective of the study was to assess the safety of apatinib mesylate administered in adult healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years of age, male or female, each gender should be more than 1/4 of the whole sample size.
2. The weight of male subject ≥50kg, weight of female subject ≥45kg, 19≤BMI≤28kg/m2
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG;
4. Agree to take approved method of contraception during the clinical trail and 8 weeks after the last dose of apatinib. Female subject should be negative in the pregnancy test;
5. Able to comprehend and willing to sign an informed consent form (ICF)

Exclusion Criteria:

1. History of drug allergy, or allergic to apatinib or ingredients;
2. Drinking 14 units of alcohol per week within 6 months prior dosing(1 unit = 360 mL of beer, or 150mL of wine) ;
3. Take any prescription or traditional Chinese medicines within four weeks prior dosing; take any over-the-counter medication, vitamin products within two weeks before dosing;
4. Take any clinical trial drugs within 3 months prior dosing;
5. Participate in blood donation within 3 months before screening and donate blood volume ≥400mL or blood loss ≥400mL, or receive blood transfusion; or donate blood volume≥200mL or blood loss ≥200mL within 1 month prior dosing.
6. Combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive) or combined with syphilis infection;
7. Anyone who refuse to stop ingest foods or drinks containing caffeine, xanthine or alcohol from 48 hours before dosing to the end of the study;
8. Anyone who refuse to stop ingesting grapefruit or grapefruit-containing products from 7 days before dosing to the end of the study;
9. The investigator believes that the subjects are not eligible to participate in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Cmax | Time Frame: Day 1: 0-72 hours; Day5: 0-72 hours;Day9:0-72hours
  Maximum Observed Plasma Concentration for apatinib [ Time Frame: Day 1: 0-72 hours; Day5: 0-72 hours;Day9:0-72hours ]
AUC0-t | Time Frame: Day 1: 0-72 hours; Day5: 0-72 hours;Day9:0-72hours
  Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration for apatinib
AUC0-inf | Time Frame: Day 1: 0-72 hours; Day5: 0-72 hours;Day9:0-72hours
  Area Under the Plasma Concentration-time Curve from Time 0 to Infinite Time for apatinib

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided